CLINICAL TRIAL: NCT03721913
Title: Efficacy of Participation-based Intervention on Community Participation and Parent Empowerment for Children With Autism Spectrum Disorder
Brief Title: Participation-based Intervention on Community Participation and Parent Empowerment for Children With ASD
Acronym: PBI-ASD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Chang Gung University (Other)
Collaborators: Chang Gung Memorial Hospital (Other)
Responsible Party: Principal Investigator, Lin-Ju Kang, Assistant Professor, Chang Gung University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 201800429A3
Record Dates: First submitted 2018-10-22; First posted 2018-10-26 (Actual); Last update posted 2022-08-26 (Actual); Status verified 2022-08

CONDITIONS: Autism Spectrum Disorder
Keywords: Autism; participation-based intervention; community participation; family empowerment; randomized controlled trial
MeSH Terms: conditions — Autism Spectrum Disorder; Autistic Disorder

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: Outcomes assessor will be masked for assessments of family empowerment
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention group (Experimental): The participation-based intervention is a goal-orientated, family-centered, and self-determined approach that emphasize on solution strategies based on child and family-selected goals. Intervention strategies will be formed by analyzing the strength and needs of child, family, and environment, and implemented by collaboration between family and interventionists.
  Interventions: Other: participation-based intervention
- Control group (No Intervention): The control group will not receive the intervention during the study.

INTERVENTIONS:
Other: participation-based intervention — The participation-based intervention is a goal-orientated, family-centered, and self-determined approach that emphasize on solution strategies based on child and family-selected goals. Intervention strategies will be formed by analyzing the strength and needs of child, family, and environment, and implemented by collaboration between family and interventionists.
  Arms: Intervention group

SUMMARY:
Community participation of children with ASD is affected by child (including body function and personal factors), family and environmental factors. This study proposes an innovative Participation-based intervention based on the principles of self-determined, family-centered, strength-based, and solution-focused approaches. This intervention targets on promoting children's community participation, and forms solution strategies from analyzing the strength and needs of child, family, and environment. The aim of this study is to investigate the efficacy of participation-based intervention on community participation and family empowerment for children with ASD 6-10 years of age.

DETAILED DESCRIPTION:
Children with Autism Spectrum Disorder (ASD) have social interaction and communication disorders, restricted interests and repetitive behaviors, which may further restrict daily activities and participation. Participation of children with ASD often are more restricted in the community than at home and school, due to problems such as environmental barriers and resources inadequacy. Research showed that school-age children with ASD participated less in social, leisure and sports activities than children with typical development, thus may result in loneness or social isolation and impact on long-term physical and psychological health.

Community participation of children with ASD is affected by child (including body function and personal factors), family and environmental factors. This study proposes an innovative Participation-based intervention based on the principles of self-determined, family-centered, strength-based, and solution-focused approaches. This intervention targets on promoting children's community participation, and forms solution strategies from analyzing the strength and needs of child, family, and environment. The aim of this study is to investigate the efficacy of participation-based intervention on community participation and family empowerment for children with ASD 6-10 years of age.

This study is proposed as a 2-year project that will use a stratified randomized controlled trial design to examine the efficacy of participation-based intervention (experimental group) in comparison to no additional intervention (control group). The study period includes 12-week intervention phase and 12-week follow-up phase, and 3 outcome measures: pre-test, post-test, and follow-up. The primary outcomes are children's community participation, the secondary outcomes are parental empowerment, family quality of life, and satisfaction with partnerships. This study will have great impact on promoting collaboration among child, family and therapists, and supporting full inclusion in society of children with ASD and their families.

ELIGIBILITY:
Inclusion Criteria:

* Children are elementary school students between the ages of 6 and 10
* Diagnosed with Autism spectrum disorder by DSM-V with a medical certificate, and reached the cut-off score (7 points) of Autism Behavior Checklist-Taiwan version(ABC-T).
* Children have an IQ of at least 70 (as measured by Wechsler Intelligence Scale for Children).
* Parents agree to participate in this study and sign the consent form.
* Children over 7 years should provide written consent form.

Exclusion Criteria:

* Children with unstable physical conditions within 3 months, such as cancer, having surgery, infection, or other active medical conditions.
* Children have known genetic conditions (e.g., Down syndrome, Fragile X Syndrome).
* Children have diagnosis associated with physical disability (e.g. cerebral palsy, congenital malformations, or musculoskeletal disorders)
* Children have significant sensory impairments such as visual or hearing impairments.

Ages: 6 Years to 10 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 24 (Actual)
Dates: Start 2018-10-23 (Actual); Primary Completion 2020-12-30 (Actual); Study Completion 2020-12-30 (Actual)

PRIMARY OUTCOMES:
Change in the Canadian Occupational Performance Measure (COPM) performance and satisfaction scores | From baseline to post-intervention at 12 weeks and follow-up at 24 weeks
  The COPM is a measure for identifying children's participation problems and prioritizing the goals. The parents will be asked to use a 10-point rating scales (1-10: higher scores indicating better performance and higher satisfaction) to rate their perception of performance and satisfaction of the goals.
Change in the Goal Attainment Scaling (GAS) scores | From baseline to post-intervention at 12 weeks and follow-up at 24 weeks
  The GAS is a measure for evaluating the goal attainment. It is a five level scale ranged from -2 to +2 where -2 represented the level of performance before intervention, 0 the expected level of attainment after intervention and +2 represented a level of attainment that exceeded expectations.

SECONDARY OUTCOMES:
Parent Empowerment and Efficacy Measure (PEEM) | Baseline, post-intervention at 12 weeks and follow-up at 24 weeks
  The PEEM is a 20-item questionnaire designed to measure parent functioning. The parents will be asked to use a 10-point scale to indicate how well each statement captures the way they feel about themselves in relation to their role as parent. A rating of 1 is used to indicate that the statement is a poor match for the way they feel and sounds nothing like them. A rating of 10 indicates that the statement is a perfect match and describes exactly how they feel. The total possible score ranges from 20 to 200.
Family Quality of Life (FaQoL) | Baseline, post-intervention at 12 weeks and follow-up at 24 weeks
  The FaQoL(McWilliam, 2011) is a 40-item questionnaire rate on a 5-point scale (1-poor to 5-excellent) for parents to rate their perception of satisfaction.
Chinese version of Family-Professional Partnership Scale (FPPS-P-C) | post-intervention at 12 weeks and follow-up at 24 weeks
  (only for the intervention groups) The FPPS-P-C is a 18-item scale for assessing parents' perceptions of the importance of and their satisfaction with family-professional partnerships. The parents will be asked to indicate how important each item was for their partnership with a professional serving their child using a 5-point scale, ranging from 1 (not at all important) to 5 (very important).

CONTACTS AND LOCATIONS:
Overall Officials: Lin-Ju Kang, PhD, Principal Investigator — Chang Gung University
Locations (1):
- Chang Gung University, Taoyuan District, Taiwan